CLINICAL TRIAL: NCT05719571
Title: Measurement of Maximal Oxygen Uptake (VO2max) Using Mankato Submaximal Exercise Test in Young Adults
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00777 Komal
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* To measure the maximal oxygen uptake (VO2max) using Mankato Submaximal Exercise test.
* To correlate 'true' VO2max with Modified Bruce protocol and Mankato Submaximal Exercise Test.

DETAILED DESCRIPTION:
First of all, 'true' VO2max of all subjects was calculated using non-exercise regression equation and one mile walk test. Variables used for the VO2max regression equation included BMI, age (years), gender (Male=1, Female=0) and physical activity rating scale. On the same visit, the subjects also performed one mile walk test. After the completion of test, pulse rate of subjects was calculated in beats per minute. The VO2max after the test was measured using the VO2max aerobic capacity calculator. Variables required were age, gender, weight, total time taken to complete test and pulse rate at test completion.

'True' VO2max accepted was the highest value obtained from non-exercise regression equation and one mile walk test On the 2nd visit, the participants performed Modified Bruce Submaximal Exercise test depending upon their fitness level and Mankato Submaximal Exercise test in counter balanced order with 30 minutes rest in between

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged between 18-35 years
* Individuals with normal BMI i.e. 18.5-24.9
* Individuals with positive cardiovascular family history

Exclusion Criteria:

* Subjects with any known cardiovascular & pulmonary disease
* Subjects addicted to caffeine/ smoking
* Subjects with any neuromuscular disability/deformity

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: study design was Analytical (Correlational) study design. During the first visit, First of all, 'true' VO2max of all subjects was calculated using non-exercise regression equation and one mile walk test.
  On the 2nd visit, the participants performed Modified Bruce Submaximal Exercise test depending upon their fitness level and Mankato Submaximal Exercise test in counter balanced order with 30 minutes rest in between.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
PAR Scale | 1 Day
  PAR scale is a self reported physical activity rating scale used for a healthy population. It describes the physical activity level of an individual from the last 6 months. It consists of scale from 0-15.
Pulse Rate | 1 Day
  Beat per minute it is measured through Pulse Oximeter
Oxygen Saturation | 1 Day
  It is measured in percentage of Oxygen in tissue, measured through Pulse oximeter
One Mile Walk Test | 1 Day
  One mile walk test is also termed as Rockport Fitness Walking Test. The subject walk distance of 1 mile and take record of the time took to cover that distance. The subject's pulse rate is taken after the completion of test by pulse oximeter
VO2max Aerobic Capacity Calculator | 1 Day
  VO2max aerobic capacity calculator is an online calculator used to measure VO2max. It calculates VO2max using the four most common methods which include, VO2max based on resting heart rate, VO2max based on one mile walk test, VO2max based on three minute step test and VO2max based on 1.5 mile walk or run test
Non-Exercise Regression Equation | 1 Day
  Non-exercise regression equation is used for measuring VO2max based on non-exercise data. The variables required for the following equation are PAR scale, age, BMI and gender.
  VO2max (ml/kg/min) = 56.363 + 1.921 × PAR - 0.381 × Age - 0.754 × BMI + 10.987 × Gender
Metabolic Equations | 1 Day
  ACSM metabolic equations are used for measuring VO2max. These metabolic equations are mentioned in ACSM's Guidelines for Exercise Testing and Prescription 2018. Following metabolic equations are used:
  * Speak (m.min-1) = (VO2max - 3.5) ∕0.2
  * Running VO2max (ml/kg/min) = (0.1 × speed) + (1.8 × speed × grade) + 3.5
  * Walking VO2max (ml/kg/min) = (0.2 × speed) + (0.9 × speed × grade) + 3.5
Modified Bruce protocol | 1 Day
  Modified Bruce protocol is a treadmill protocol and modified form of Bruce protocol with decreased increment in initial stages and then increasing the slope progressively. Following are the Modified Bruce protocol stages:
  Stage 0 = 1.7 mph at 0% Grade Stage 0.5 = 1.7 mph at 5% Grade Stage 1 = 1.7 mph at 10% Grade Stage 2 = 2.5 mph at 12% Grade Stage 3 = 3.4 mph at 14% Grade Stage 4 = 4.2 mph at 16% Grade Stage 5 = 5.0 mph at 18% Grade Stage 6 = 5.5 mph at 20% Grade Stage 7 = 6.0 mph at 22% Grade Stage 8 = 6.5 mph at 24% Grade

CONTACTS AND LOCATIONS:
Overall Officials: Anam Aftab, PPDPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Pakistan, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No